CLINICAL TRIAL: NCT03183960
Title: Stroke - 65 Plus. Continued Active Life. A Randomised Controlled Trial of the Effect of a Novel Self-management Intervention Supporting Older Adults After Stroke
Brief Title: Stroke - 65 Plus. Continued Active Life.
Acronym: Stroke65+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Hanne Pallesen, Physiotherapist, PhD. Head of Clinical Physiotherapy Research, at Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Denmark, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: JutlandRH54962
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Self-management; Quality of Life
Keywords: Self-management; Quality of Life; Self-efficacy; Support; Stroke; Older adults
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentor (Experimental): An independent centralized randomization database will provide allocation concealed to the involved clinicians and assessors. A stratified block randomization of severity of impairment will be performed within each rehabilitation hospital
  Interventions: Behavioral: Mentor
- Traditional rehabilitation (Active Comparator): An independent centralized randomization database will provide allocation concealed to the involved clinicians and assessors. A stratified block randomization of severity of impairment will be performed within each rehabilitation hospital
  Interventions: Behavioral: Mentor

INTERVENTIONS:
Behavioral: Mentor — Traditional rehabilitation.
  Other Names: Self-mangement

SUMMARY:
Since august 2016, the researchers at a highly specialized neurorehabilitation hospital in a Danish region with 1.2 inhabitants have in cooperation with health professionals from a specialized neurorehabilitation in a Danish municipality with 336,000 inhabitants, worked through and is still working with an iterative process in the development of a novel self-management support intervention for elderly stroke individuals.The intervention is going to be implemented into the second phase- a randomized clinical controlled trial (RCT) in the project named 'Stroke - 65 plus. Continued active life'.

DETAILED DESCRIPTION:
Background: Elderly adults represent the majority of stroke cases worldwide. Sequelae after a stroke causes the stroke individuals to live a more isolated life 5 years after the stroke. This makes the stroke individuals an especially vulnerable group of elderly people regarding social reintegration. Reintegration into the community post-stroke depends highly on support from the family. However, the stroke individual's closest relatives are at risk of developing anxiety and depression.

The aim of this study is to investigate the effect of a novel self-management intervention supporting older adults after stroke

Methods/Design: Randomized controlled observer-blind trial. More than sixty stroke survivors over 65 years will two weeks before leaving a rehabilitation hospital be randomized to either a group receiving conventional rehabilitation (control) or a novel self-management intervention addition to standard rehabilitation.

During a period of 6 months the patients will be offered additional 6-8 sessions of self-management intervention of 45-60 minutes duration by a physiotherapist or an occupational therapist.

Study outcome measurements: Stroke Self-efficacy questionnaire, Stroke Specific Quality of Life Scale and Impact on participation and Autonomy and activity by accelerometers will be evaluated at baseline, three and nine months post hospital treatment.

Patient, informal caregiver and therapist satisfaction will be with examined with questionnaires and interviews.

Discussion: Self-management interventions are promising tools for rehabilitation of self-efficacy, quality of life as well as participation and autonomy. The introduction of novel self management intervention in combination with traditional physical and occupational therapy may enhance recovery after stroke, quality of life and burden on relatives. Stroke 65+ trial will provide further evidence of self management strategies to clinicians, patients and health economists.

ELIGIBILITY:
Inclusion Criteria:

* stroke survivors with rehabilitation needs discharge from rehabilitation hospital to home

Exclusion Criteria:

* do not understand danish Montreal Cognitive assessment (MOCA) below 20

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Stroke Self-efficacy questionnaire | Measured at baseline, 3 and 9 months post discharged from rehabilitation hospital
  Change of Self-efficacy

SECONDARY OUTCOMES:
Impact on participation and Autonomy Questionnaire | Measured 3 and 9 months post discharged from rehabilitation hospital
  Change of Impact on participation and Autonomy
Stroke Specific Quality of Life Scale Questionnaire(short version) | Measured at baseline, 3 and 9 months post discharged from rehabilitation hospital
  Change of Specific Quality of Life

OTHER OUTCOMES:
Activity (accelerometers) | Measured at baseline, 3 and 9 months post discharged from rehabilitation hospital
  Change of activity
Caregiver Burden Scale | Measured at baseline, 3 and 9 months post discharged from rehabilitation hospital
  Change of caregivers burden

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Pallesen, Post Doc, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (2):
- Denmark (2):
  - Region Hospital Hammel Neurocentre, Hammel, Jutland
  - Region Hospital Hammmel Neurorehabilitation, Hammel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pallesen H, Pedersen SKS, Sorensen SL, Naess-Schmidt ET, Brunner I, Nielsen JF, Kjeldsen SS. "Stroke - 65 plus. Continued active life." A randomized controlled trial of a self-management neurorehabilitation intervention for elderly people after stroke. Disabil Rehabil. 2025 Jan;47(1):104-113. doi: 10.1080/09638288.2024.2338190. Epub 2024 Apr 8. PMID 38587056
- [Derived] Pedersen SKS, Pallesen H. Stroke self-efficacy questionnaire - Denmark (SSEQ-DK): test-retest of the Danish version. Top Stroke Rehabil. 2023 Mar;30(2):193-202. doi: 10.1080/10749357.2021.2016097. Epub 2022 Jan 7. PMID 34994306
- [Derived] Sorensen SL, Pedersen SKS, Pallesen H. Social psychological mechanisms and processes in a novel, health professional-led, self-management intervention for older stroke individuals: a synthesis and phenomenological study. BMC Health Serv Res. 2019 May 22;19(1):320. doi: 10.1186/s12913-019-4150-x. PMID 31113442
- [Derived] Pallesen H, Naess-Schmidt ET, Kjeldsen SS, Pedersen SKS, Sorensen SL, Brunner I, Nielsen JF. "Stroke - 65 Plus. Continued Active Life": a study protocol for a randomized controlled cross-sectoral trial of the effect of a novel self-management intervention to support elderly people after stroke. Trials. 2018 Nov 19;19(1):639. doi: 10.1186/s13063-018-2961-4. PMID 30454014